CLINICAL TRIAL: NCT04277390
Title: Evidence Linking the Role of Viruses, Bacteria and Placental MIR155 in Chronic Periodontitis and Preeclampsia- A Genetic Microbiological Study
Brief Title: microRNA 155 Levels and Periodontal Microflora (Bacteria and Virus) in Preeclampsia.
Status: Completed | Type: Observational
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Professor, PhD guide, Director of Post Graduate Studies, Meenakshi Ammal Dental College and Hospital
Other Study IDs: NDC/staff/2015-16/EC/2015
Record Dates: First submitted 2020-02-12; First posted 2020-02-20 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Preeclampsia; Chronic Periodontitis
Keywords: periodontal microflora, preeclampsia
MeSH Terms: conditions — Pre-Eclampsia; Chronic Periodontitis | interventions — imidazole mustard; Biomarkers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — subgingival plaque samples and placental tissue samples were obtained. DNA was isolated and then subjected to RTPCR for microbial identification and estimation of MIR155 levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Controls: 145 systemically and periodontally healthy pregnant women Subgingival samples and placental tissue samples(postpartum) were collected for microbial analysis and check for the levels of MIR155.
  Interventions: Other: clinical intervention for microbial analysis and MIR155 as biomarker
- Group A: Group A-100 Systemically healthy pregnant women with chronic periodontitis.
  Subgingival samples and placental tissue samples(postpartum) were collected for microbial analysis and check for the levels of MIR155.
  Interventions: Other: clinical intervention for microbial analysis and MIR155 as biomarker
- Group B: Group B- 100 Preeclamptic pregnant women with chronic periodontitis. Subgingival samples and placental tissue samples(postpartum) were collected for microbial analysis and check for the levels of MIR155.
  Interventions: Other: clinical intervention for microbial analysis and MIR155 as biomarker
- Group C: Group C-100 Preeclamptic pregnant women without chronic periodontitis. Subgingival samples and placental tissue samples(postpartum) were collected for microbial analysis and check for the levels of MIR155.
  Interventions: Other: clinical intervention for microbial analysis and MIR155 as biomarker

INTERVENTIONS:
Other: clinical intervention for microbial analysis and MIR155 as biomarker — Subgingival plaque was collected with sterile curette and placental tissue sample(postpartum with surgical blade with the help of gynecologist. all the samples were subjected to RTPCR for analysis of microorganisms likeTannerella forsythia(Tf), Treponema denticola(Td), Porphyromonas gingivalis(Pg), Prevotella intermedia(Pi), Fusobacterium nucleatum(Fn). Herpes Simplex Virus(HSV), Ebstein Barr Virus(EBV), Human Cytomegalovirus(HCMV). and MIR155 levels were also estimated

SUMMARY:
Preeclamptic women with and without chronic periodontitis were recruited for the study. Subgingival plaque samples and placental tissue samples(postpartum) were obtained from the participants for the microbial analysis(bacteria, viruses) and MIR155 levels and comparison was done among groups. this study was designed in order to evaluate the role of periodontal microorganisms in preeclampsia and to find compare the MIR155 levels among participants, so as to check its importance as a biomarker for inflammatory disease like preeclampsia.

DETAILED DESCRIPTION:
Four hundred forty five pregnant women, aged 18-35 yrs were selected and were divided into four groups. Controls- 145 systemically and periodontally healthy, Group A-100 Systemically healthy women with chronic periodontitis, Group B- 100 Preeclamptic women with chronic periodontitis, Group C-100 Preeclamptic women without chronic periodontitis. Age, BMI, Socioeconomic status and periodontal parameters such as plaque index(PI), bleeding on probing(BOP), probing pocket dept(PPD), clinical attachment level(CAL) were recorded. Subgingival plaque and placental tissues (postpartum) were collected and assessed for periodontal pathogens such as Tannerella forsythia(Tf), Treponema denticola(Td), Porphyromonas gingivalis(Pg), Prevotella intermedia(Pi), Fusobacterium nucleatum(Fn). Herpes Simplex Virus(HSV), Ebstein Barr Virus(EBV), Human Cytomegalovirus(HCMV). microRNA155 levels were also assessed and compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women within the age group of 18-35 years with single gestation, having ≥ 20 natural teeth, who did not receive periodontal treatment in last six months and willing to participate in the study were included for the investigation.

Exclusion Criteria:

* Pregnant women with current use of any form of tobacco, history of alcohol consumption and systemic medications were excluded from the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Controls- 145 systemically and periodontally healthy pregnant women, Group A-100 Systemically healthy pregnant women with chronic periodontitis, Group B- 100 Preeclamptic pregnant women with chronic periodontitis, Group C-100 Preeclamptic pregnant women without chronic periodontitis.
Sampling Method: Non-Probability Sample
Enrollment: 445 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
Viruses, Bacteria and placental mir155 in Chronic Periodontitis and Preeclampsia | it took approximately 15 minutes to collect samples for DNA extraction.
  Viruses, Bacteria and placental mir155 were assessed in Chronic Periodontitis and Preeclamptic pregnant women.

CONTACTS AND LOCATIONS:
Overall Officials: Jaideep Mahendra, MDS, PhD, Study Director — Meenakshi Ammal Dental College
Locations (1):
- Swetha Tanneeru, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barak S, Oettinger-Barak O, Machtei EE, Sprecher H, Ohel G. Evidence of periopathogenic microorganisms in placentas of women with preeclampsia. J Periodontol. 2007 Apr;78(4):670-6. doi: 10.1902/jop.2007.060362. PMID 17397314
- [Background] Jaiman G, Nayak PA, Sharma S, Nagpal K. Maternal periodontal disease and preeclampsia in Jaipur population. J Indian Soc Periodontol. 2018 Jan-Feb;22(1):50-54. doi: 10.4103/jisp.jisp_363_15. PMID 29568173
- [Background] Mahendra J, Parthiban PS, Mahendra L, Balakrishnan A, Shanmugam S, Junaid M, Romanos GE. Evidence Linking the Role of Placental Expressions of Peroxisome Proliferator-Activated Receptor-gamma and Nuclear Factor-Kappa B in the Pathogenesis of Preeclampsia Associated With Periodontitis. J Periodontol. 2016 Aug;87(8):962-70. doi: 10.1902/jop.2016.150677. Epub 2016 May 13. PMID 27177289
- [Background] Reddy BV, Tanneeru S, Chava VK. The effect of phase-I periodontal therapy on pregnancy outcome in chronic periodontitis patients. J Obstet Gynaecol. 2014 Jan;34(1):29-32. doi: 10.3109/01443615.2013.829029. PMID 24359045